CLINICAL TRIAL: NCT01435824
Title: Bioavailability of Amoxicillin Dissolved in Human Milk: An Adult Volunteer Study as a First Step Towards Defining Drug Doses for Infants
Brief Title: Bioavailability of Amoxicillin Dissolved in Human Milk
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Shinya Ito, Division Head, Clinical Pharmacology and Toxicology, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1000021187
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Healthy
Keywords: healthy adult volunteers; comparative bioavailability; amoxicillin; breast milk; Amoxicillin Bioavailability in breast milk

STUDY DESIGN:
Intervention Model Description: Participants underwent 2 arms in a cross-over design: 1 ) amoxicillin disolved in water; and 2) amoxicillin dissolved in human milk. The order of the 2 arms were randomized.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Water as a vehicle of amoxicillin (Active Comparator): Amoxicillin 500 mg was dissolved in 10 ml water and orally administered in a fasting state.
  Interventions: Drug: Water-dissolved amoxicillin
- Human milk as a vehicle of amoxicillin (Experimental): Amoxicillin 500 mg was dissolved in 10 ml human milk and orally administered in a fasting state.
  Interventions: Drug: Human milk-dissolved amoxicillin

INTERVENTIONS:
Drug: Human milk-dissolved amoxicillin — An amoxicillin suspension bottle containing 5 grams of amoxicillin (powder) will be resuspended in 60 ml of breast milk to have 100mL of a 50mg/mL suspension.
  Other Names: Novamoxin 250 from Novopharm, Toronto, Canada: Lot#35422063A; Frozen human milk was obtained from the Mother's Milk Bank of Ohio (USA)
  Arms: Human milk as a vehicle of amoxicillin
Drug: Water-dissolved amoxicillin — An amoxicillin suspension bottle containing 5 grams of amoxicillin (powder) will be resuspended in 60 ml of water to have 100mL of a 50mg/mL suspension.
  Other Names: Novamoxin 250 from Novopharm, Toronto, Canada: Lot#35422063A
  Arms: Water as a vehicle of amoxicillin

SUMMARY:
The investigators propose to study amoxicillin absorption in a 2-stage program that will progressively produce, for the first time, information leading to pediatric pharmacology recommendations for the administration to children of amoxicillin dissolved in human milk. The investigators study will enroll adult volunteers as number of blood extractions, volume of blood required and subject availability, among other issues, generate a number of ethical and logistical constraints that make it almost impossible to carry such an intensive sampling study in infants.

DETAILED DESCRIPTION:
As recommended by the Expert Committee on Selection and Use of Essential Medicines, WHO (http://www.who.int/selection_medicines/committees/en/index.html), oral solid formulations are the preferred forms of medicines for children, especially in developing countries, because of relatively inexpensive and less complicated manufacturing, transporting and storage processes. Whereas solid dosage forms are advantageous in these pharmaceutical logistics, administering solid formulations to infants and children is a challenging issue. Dissolving medicines in water may be acceptable, but safety of drinking water for infants in developing countries and water solubility of the drug itself are major concerns. These challenges are exemplified in the treatment of infectious diseases and diarrhea in infants. Commonly used drugs for infants in low income settings include antibiotics such as amoxicillin. Expert sources have suggested that drug administration in breast milk may be effective. However, little data is currently available to support the recommendation to administer medications dissolved in breast milk to infants.

The second stage of the project will use the information obtained from the first stage, combined with pre-existing data, to define a rational dosing schedule of the target drug dissolved in human milk for young children, using population PK modeling and simulation. This is a study in silico.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers (>18 and <60 years old)
2. An approximate 50% of the volunteers will be female
3. Body mass index (BMI) within 18.5 to 29.9 kg/m2
4. Healthy according to medical history, vital signs and a brief physical examination as determined by the principal investigator/Sub-investigators.
5. Systolic blood pressure between 100-140 mmHg, inclusive and diastolic blood pressure between 60-90 mmHg, inclusive, and heart rate between 50-100 bpm, unless deemed not clinically significant by the principal investigator/Sub- investigators.
6. Capable of giving written informed consent prior to receiving study medication
7. Smoking is not an exclusion criterion but we will identify smokers.
8. Female participants will be required to fulfill at least one of the following:

   * Agree to avoid pregnancy and use medically acceptable method of contraception from at least 30 days prior to the study, during the study, and until 30 days after to the study has ended (last study procedure). Medically acceptable methods of contraception include hormonal patch, implant or injection intrauterine device, or double barrier method (condom with foam or vaginal spermicidal suppository, diaphragm with spermicidal). Complete abstinence alone can be used as a method of contraception. Oral contraceptives prior to the study are acceptable as a method of contraception, but an alternative method of contraception will be required during the study and after the study has ended.
   * Be surgically sterile for a minimum of 6 months
   * Post menopausal for a minimum of 1 year.

Exclusion Criteria:

1. Known history of any clinically significant hepatic (e.g. hepatic necrosis, jaundice, hepatobiliary disease), renal, gastrointestinal (e.g. peptic ulcer), cardiovascular (e.g. angina, myocardial infarction), cerebrovascular, pulmonary, endocrine (e.g. diabetes, hypophosphatemia), immunological, musculoskeletal (e.g. rhabdomyolysis, myopathy), neurological, psychiatric, dermatological, or haematological disease or condition
2. History of any clinically significant illness within 30 days prior to dosing
3. History of any significant physical or organ abnormality
4. Known history of:

   * Alcohol abuse or dependence within one year prior to drug administration
   * Drug abuse or dependence
   * Food allergies and/or presence of any dietary restrictions
   * Severe allergic reactions (e.g. anaphylactic reactions, angioedema)
5. Participation in another clinical trial or receiving an investigational drug within 30 days of the study commencement or during the study
6. Use of any prescription medication within 14 days prior to drug administration (except for hormonal contraceptives)
7. Use of any over the counter medications )including herbal and/or dietary supplements and/or teas) within 24 hrs prior to drug administration (except for spermicidal/barrier contraceptive products)
8. Any major surgery within 6 months prior to the start of the study
9. History of allergy to amoxicillin, beta-lactams or amoxicillin excipients
10. History of allergy to milk, or severe lactose intolerance
11. Pregnancy or lactating
12. Conditions associated with malabsorption
13. Taking any form of antacids as they may increase the risk of orally transmitted viruses from human milk.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-06; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shinya Ito, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- See also: Link to published study results — http://dx.doi.org/10.1136/archdischild-2013-305151

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy young adults were enrolled. 16 individuals were assessed and randomly assigned to either "water-based first, then milk-based amoxicillin administration" or "milk-based first and then water-based administration" arms. The washout period was 1-2 weeks. The study was conducted at Hospital for Sick Children in Toronto, Canada.
Pre-assignment Details: Participants were interviewed and underwent basic vital sign checking, and filled health status questionnaire to declare lack of any significant medical conditions. Urine pregnancy tests, with consents, were performed before dosing for female participants.Wash-out period between water and human milk phases was 1-2 weeks.
Groups:
- Water-based First, Then Milk-based Administration: First, participants were orally given 10 mL of water-dissolved amoxicillin (50mg/mL) in a fasting state. A PK sampling was performed. The washout period was for 1-2 weeks and then participants underwent the milk-based administration of amoxicillin, followed by PK sampling.
- Milk-based First, and Then Water-based Drug Administration: First, participants were orally given 10 mL of human milk-dissolved amoxicillin (50mg/mL) in fasting state, followed by PK sampling. The washout period was for 1-2 weeks and then participants underwent a water-based administration if amoxicillin followed by PK sampling. .
Period: First Intervention
Arm/Group | Water-based First, Then Milk-based Administration | Milk-based First, and Then Water-based Drug Administration
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout of 1-2 Weeks
Arm/Group | Water-based First, Then Milk-based Administration | Milk-based First, and Then Water-based Drug Administration
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Water-based First, Then Milk-based Administration | Milk-based First, and Then Water-based Drug Administration
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: This study was designed as a randomized 2x2 crossover single-dose study where participants either given water-dissolved amoxicillin first or human milk-dissolved amoxicillin first switched over during period 2.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 16
Height [Mean (Standard Deviation); unit: cm] | 167.6 (12.3)
Weight [Mean (Standard Deviation); unit: kg] | 67.1 (14.3)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve to Time Infinity (AUC to Time Infinity)
Description: Amoxicillin plasma concentrations were determined by HPLC-MS/MS and AUC∞ (to time infinity) was estimated using a model-independent approach. Specifically, the log-trapezoidal method was used to calculate AUC last (AUC from time 0 to 8 h), and AUC∞ was further estimated with the elimination rate constant (Kel) of the terminal log-linear phase (β phase) of the concentration time profile extrapolating to time infinity as follows:
  AUC∞ = AUC last + [C]8h/Kel; where [C]8h is the plasma concentration at time 8 h postdose.
Time Frame: Baseline, 0.25, 0.5, 1, 1.5, 3, 4 and 8 hours after dosing
Measure: Mean (Standard Deviation); unit: mcg*min/mL
Arm/Group | Water as a Vehicle of Amoxicillin | Human Milk as a Vehicle of Amoxicillin
Number analyzed (Participants) | 16 | 16
mcg*min/mL | 1394.1 (256.1) | 1477.2 (260.7)
Statistical Analysis 1: Comparison: Water as a Vehicle of Amoxicillin vs Human Milk as a Vehicle of Amoxicillin; A 2x2 crossover design was chosen to examine bioequivalence of milk-based amoxicillin preparation, based on the FDA-recommended design for bioavailability studies. The recommendation suggests that 12 subjects is the minimum number of subjects acceptable for this type of design. We have decided to enrol 16 subjects to account for problems or attrition; Test type: Equivalence — Bioequivalence is assessed by means of ratios of AUC, Cmax and Tmax between the comparison group and the reference group. According to a common regulatory definition, the comparison preparation (human milk-dissolved amoxicillin in this project) is considered bioequivalent to a standard preparation (water dissolved) if 90% CIs of these ratios between the two preparations for Cmax, Tmax, AUClast and AUC∞ are within a range between 0.80 and 1.25; mean %ratio and 90% confidence interval = 106.1, 90% CI 2-sided [97.5 to 115.4]

2. Primary Outcome: Area Under the Curve to 8h (AUC Last)
Description: Amoxicillin plasma concentrations were determined by HPLC-MS/MS and PK parameters were estimated using a model-independent approach. Specifically, the log-trapezoidal method was used to calculate AUC last (AUC from time 0 to 8 h).
Time Frame: Baseline, 0.25, 0.5, 1, 1.5, 3, 4 and 8 hours after dosing
Measure: Mean (Standard Deviation); unit: mcg*min/mL
Arm/Group | Water as a Vehicle of Amoxicillin | Human Milk as a Vehicle of Amoxicillin
Number analyzed (Participants) | 16 | 16
mcg*min/mL | 1355.8 (254.2) | 1435.0 (241.7)
Statistical Analysis 1: Comparison: Water as a Vehicle of Amoxicillin vs Human Milk as a Vehicle of Amoxicillin; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; mean %ratio and 90% confidence interval = 106.2, 90% CI 2-sided [97.5 to 115.7]

3. Primary Outcome: Cmax
Description: A maximum plasma concentration of amoxicillin within the time frame of a dosing
Time Frame: 0, 0.25, 0.5, 1, 1.5, 3, 4 and 8 hours after dosing
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Water as a Vehicle of Amoxicillin | Human Milk as a Vehicle of Amoxicillin
Number analyzed (Participants) | 16 | 16
ng/ml | 8653.8 (2217.6) | 8690.6 (1972.4)
Statistical Analysis 1: Comparison: Water as a Vehicle of Amoxicillin vs Human Milk as a Vehicle of Amoxicillin; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; mean %ratio and 90% confidence interval = 101.3, 90% CI 2-sided [89.4 to 114.9]

4. Primary Outcome: Tmax
Description: Time to reach Cmax after administration
Time Frame: Data points were taken at 0, 0.25, 0.5, 1, 1.5, 3, 4 and 8 hours after dosing.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Water as a Vehicle of Amoxicillin | Human Milk as a Vehicle of Amoxicillin
Number analyzed (Participants) | 16 | 16
min | 101.3 (52.4) | 106.9 (49.0)
Statistical Analysis 1: Comparison: Water as a Vehicle of Amoxicillin vs Human Milk as a Vehicle of Amoxicillin; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; mean %ratio and 90% confidence interval = 107.9, 90% CI 2-sided [84.5 to 137.8]

5. Secondary Outcome: Elimination Half-life
Description: Elimination rate constant (Kel) was estimated from the terminal log-linear phase of the concentration-time profiles. Then, elimination half-life was calculated as follows: ln2/Kel.
Time Frame: Data points were taken at 0, 0.25, 0.5, 1, 1.5, 3, 4 and 8 hours after dosing.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Water as a Vehicle of Amoxicillin | Human Milk as a Vehicle of Amoxicillin
Number analyzed (Participants) | 16 | 16
min | 77.7 (17) | 76.1 (11.7)

6. Secondary Outcome: Clearance/F
Description: The log-trapezoidal method was used to calculate AUC last (AUC from time 0 to 8 h), and AUC∞ was estimated using an elimination rate constant (Kel) of the terminal log-linear phase (β phase) of the concentration time profile extrapolating to time infinity. Then, CL/F was derived from Dose/AUC∞. F is bioavailability, which cannot be determined in this study, and therefore, we estimate CL/F, but not CL itself.
Time Frame: Data points were taken at 0, 0.25, 0.5, 1, 1.5, 3, 4 and 8 hours after dosing.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Water as a Vehicle of Amoxicillin | Human Milk as a Vehicle of Amoxicillin
Number analyzed (Participants) | 16 | 16
ml/kg/min | 5.63 (1.05) | 5.34 (1.22)

7. Secondary Outcome: Volume of Distribution/F
Description: It was estimated from (Clearance/F)/Kel. Elimination rate constant (Kel) was estimated from the terminal log-linear phase of the concentration-time profiles. Then, elimination half-life was calculated as follows: ln2/Kel.
Time Frame: Data points were taken at 0, 0.25, 0.5, 1, 1.5, 3, 4 and 8 hours after dosing.
Measure: Mean (Standard Deviation); unit: l/kg
Arm/Group | Water as a Vehicle of Amoxicillin | Human Milk as a Vehicle of Amoxicillin
Number analyzed (Participants) | 16 | 16
l/kg | 0.63 (0.18) | 0.59 (0.16)

ADVERSE EVENTS:
Time Frame: 1 week
Groups:
- Water-based Amoxicillin Administration: Amoxicillin was dissolved in water and administered for PK sampling.
- Human Milk-based Amoxicillin Administration: Amoxicillin was dissolved in human milk and administered for PK sampling.
Arm/Group | Water-based Amoxicillin Administration | Human Milk-based Amoxicillin Administration
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
Participants ingested amoxicillin dissolved in 10 mL of milk or water. We cannot rule out that larger volumes of milk can change absorption profile of the drug.

PK parameters in adults may be different from those reported in neonates and infants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes